CLINICAL TRIAL: NCT00344981
Title: A Study to Probe The Safety And Durability of Tenofovir And a Cell Cycle Agent to Maintain Viral Suppression
Brief Title: Safety and Durability ofTenofovir and a Cell Cycle Agent for Viral Suppression
Acronym: HADIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Dr. Robert R. Redfield, Institute of Human Virology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-22407
Record Dates: First submitted 2006-06-23; First posted 2006-06-27 (Estimated); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: HIV Infections; AIDS
Keywords: Cell Cycle Agents
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Tenofovir; Hydroxyurea

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Tenofovir — Half of the 20 volunteers will be randomized to the Tenofovir 300 mg qd/Hydroxyurea 500mg qd arm and those subjects will have Hydroxyurea added to their current screening regimen for 4 weeks prior to de-intensifying to Hydroxyurea and Tenofovir.
  Other Names: Viread
Drug: Hydroxyurea — Half of the 20 volunteers will be randomized to the Tenofovir 300 mg qd/Hydroxyurea 500mg qd arm and those subjects will have Hydroxyurea added to their current screening regimen for 4 weeks prior to de-intensifying to Hydroxyurea and Tenofovir. Volunteers will continue on this regimen for 48 weeks. Patients will be monitored for immunological and virological parameters as well as the incidence of toxicity and side effects during the study. If a patient's viral load reaches >400 copies/ml on 3 consecutive measurements over a 6 week period, they will be terminated from the study and started back on their HAART.
  Other Names: Hydrea

SUMMARY:
Study Hypothesis Evaluation of the durability of the combination Tenofovir and Hydroxyurea to maintain viral suppression below 50 copies/ml in volunteers who have achieved viral suppression on a standard HAART regimen.

DETAILED DESCRIPTION:
This is a 48 week open-label, randomized study comparing the safety and durability of a highly active de-intensified therapy (Tenofovir/Hydroxyurea) to a simplified standard of care therapy (Tenofovir plus 3TC or Emtriva plus Sustiva or Nevirapine) to maintain a durable viral suppression.

Up to 20 subjects with chronic HIV-1 infection, suppressed on highly active antiretroviral therapy, and without evidence of viral resistance will be enrolled in this study. Their present HAART therapy will be stopped.

Half of the 20 volunteers will be randomized to the Tenofovir 300 mg qd/Hydroxyurea 500mg qd arm and those subjects will have Hydroxyurea added to their current screening regimen for 4 weeks prior to de-intensifying to Hydroxyurea and Tenofovir. The other half will be randomized to Sustiva 600 mg qd or Nevirapine 200 mg twice a day); Tenofovir 300 mg qd, 3TC 300 mg qd or Emtriva 200 mg once a day. Volunteers will continue on this regimen for 48 weeks. Patients will be monitored for immunological and virological parameters as well as the incidence of toxicity and side effects during the study. If a patient's viral load reaches >400 copies/ml on 3 consecutive measurements over a 6 week period, they will be terminated from the study and started back on their HAART.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of HIV infection based on western blot testing, ELISA, or HIV viral load
2. Age greater than or equal to 18 years
3. CD4 count greater than or equal to 200c/ml.
4. On a standard HAART regimen of 2 or 3 nucleoside reverse transcriptase inhibitors and either a protease inhibitor or a nonnucleoside reverse transcriptase inhibitor or 3 nucleoside reverse transcriptase inhibitors (2-3NRTI's + PI or 2-3NRTI's +NNRTI or 3NRTI's).
5. On stable, continuous HAART regimen for greater than or equal to 3 months,
6. Viral load less than or equal to 400c/ml on all measurements in the preceding 6 months with at least 2 measurements (screening viral load can be included if needed)
7. Viral load less than or equal to 50c/ml at screening
8. Subject able to comply with the study protocol
9. Signed informed consent
10. No history of antiretroviral failure that is suspected to be from or resulted in antiretroviral resistance.

Exclusion Criteria:

1. Serious HIV related or non HIV related carcinoma requiring chemotherapy
2. Recent serious opportunistic infection, such as progressive multifocal leukoencephalopathy, CMV disease, cryptococcus meningitis, cerebral toxoplasmosis, but not excluding other infections in which successful treatment may be judged to be placed at risk if antiretroviral therapy was de intensified.
3. Known or suspected intolerance or hypersensitivity to Hydroxyurea
4. Grade 3 or higher neutropenia (using ACTG grading table)
5. Grade 2 or higher thrombocytopenia (using ACTG grading table)
6. Grade 2 or higher LFT abnormalities (using ACTG grading table)
7. History of pancreatitis, or risk factors associated with pancreatitis (more then two drinks containing alcohol/day, triglyceride levels greater than 400, and pancreatic enzymes greater then 1.5x normal)
8. Renal insufficiency (Estimated Creatinine clearance of <60ml/min.)
9. Chronic diarrhea
10. Pregnancy or breastfeeding
11. Unwillingness to use effective barrier contraception or abstinence
12. The use of systemic corticosteroids, or other systemic immunosuppressive medications; the use of cholestyramine; the use of probenecid or other inhibitors of renal tubular secretion
13. Genotypic or phenotypic testing documenting major resistance to any antiretroviral agents
14. Active substance or mental health concerns that are judged to place a significant limitation on medication adherence.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2003-06; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Loss of viral suppression during maintenance therapy, defined by 3 consecutive viral load measurements greater than 50c/ml over a 48- week period. | At any point during the 48 week study
  Viral load measurements will be done throughout the study to monitor for viral suppression

SECONDARY OUTCOMES:
Laboratory Abnormalities: Routine measurements of hematology, serum chemistry, CD4 cell count, lipid profiles, and HIV-1 viral load will be performed. Viral genotypes will be performed with failure to maintain viral suppression. | Throughout the 48 week study
  These tests will be done to monitor Safety and tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Robert R. Redfield, MD, Principal Investigator — University of Maryland, School of Medcine, Department of Infectious Disease
Locations (1):
- University of Maryland, Institute of Human Virology, Baltimore, Maryland, United States